CLINICAL TRIAL: NCT03858465
Title: Comparison of Phenylephrine and Ephedrine in the Treatment of Hemodynamic Disorders After Spinal Anesthesia in the Elderly
Acronym: HypoGer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Rafal Kowalczyk, Principal Investigator, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KB/129/2017
Record Dates: First submitted 2019-02-20; First posted 2019-02-28 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Hip Fractures; Elderly Patients; Spinal Anesthesia; Lower Limb Surgery
Keywords: Hypotension; Phenylephrine; Ephedryne
MeSH Terms: conditions — Hip Fractures; Hypotension | interventions — Ephedrine; Phenylephrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 25 mg of ephedrine (Active Comparator): participants who will receive intravenous 1,25mg/min ephedrine during 20 minutes (total dosage is 25 mg of ephedrine).
  Interventions: Drug: Ephedrine
- 0,3 mg of phenylephrine (Active Comparator): participants who will receive intravenous 0,015mg/min phenylephrine during 20 minutes (total dosage is 0,3mg of phenylephrine).
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Ephedrine — intravenous 25 mg of ephedrine
  Other Names: Ephedrinum hydrochloricum WZF Polfa Warszawa 25mg/ml
  Arms: 25 mg of ephedrine
Drug: Phenylephrine — intravenous 0,3 mg of phenylephrine
  Other Names: Phenylephrine Unimedic 10mg/ml
  Arms: 0,3 mg of phenylephrine

SUMMARY:
Spinal anesthesia is often used for lower limb surgery in elderly. Hypotension is a side effect of spinal block. In this study, intravenous ephedrine and phenylephrine will be compared with each other to prevent spinal anesthesia-induced hypotension, which is defined in absolute terms as a systolic blood pressure < 100 mmHg or in relative terms as a 20% fall of systolic blood pressure from baseline.

DETAILED DESCRIPTION:
Randomized single centre clinical randomized study will be performed on 50 participants. The inclusion criteria are participants (age more than 65 years) with proximal femoral fracture scheduled for lower limb surgery under spinal anesthesia.

The Ethics Committee approved this prospective study. Informed consent will be taken from individual subjects. Participants are randomly allocated into one of the two study groups.

Group A: participants who will receive intravenous 25 mg of ephedrine added to syringe with 50 ml 0,9% sodium chloride solution during 20 minutes. Group B: Phenylephrine 5 mg will be added to syringe with 50 ml 0,9% sodium chloride solution, participants will receive intravenous 0,3 mg of phenylephrine during 20 minutes. Randomization is achieved with the help of Random.org.

In order to reduce pain prior to spinal anesthesia an ultrasound-guided fascia iliaca block will be performed using a volume of 30 ml ropivacaine 0,2%. After skin infiltration with 3 ml of lidocaine, a 25G Pencan spinal needle will be inserted at the L3-L4 or L4-L5 vertebral interspaces. After aspirating cerebrospinal fluid, participants will receive hyperbaric bupivacaine 0.5% at 0,11 mg/cm according to the participant height. Ephedrine and phenylephrine will be given intravenous immediately after injection of bupivacaine. Impedance cardiography will be used to measure hemodynamic parameters: cardiac output, stroke volume, cardiac index, stroke index, systemic vascular resistance, systemic vascular resistance index. Heart rate, blood pressure and oxygen saturation will also be controlled. All these parameters will be measured and recorded every 5 minutes until 30 minutes after spinal anesthesia. The data will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* elderly (age more than 65 years)
* hip fracture scheduled for lower limb surgery under spinal anesthesia
* spinal anesthesia

Exclusion Criteria:

* contraindications to spinal anesthesia
* participant refusal
* age less than 65
* bradycardia (heart rate less than 60)
* participants unable to give consent or inability to communicate

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-02-24 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
blood preasure (mean arterial pressure, systolic and diastolic blood pressure) | 30 min
  parameter will be measured and recorded every 5 min after spinal anesthesia.

SECONDARY OUTCOMES:
heart rate, expressed in bpm | 30 min
  parameter will be measured using impedance cardiography and recorded every 5 min after spinal anesthesia.
cardiac output, expressed in L/min | 30 min
  parameter will be measured using impedance cardiography and recorded every 5 min after spinal anesthesia.
stroke volume, expressed in ml | 30 min
  parameter will be measured using impedance cardiography and recorded every 5 min after spinal anesthesia.
cardiac index, expressed in L/min/m2, is the ratio of cardiac output to the body surface area. | 30 min
  parameter will be measured using impedance cardiography and recorded every 5 min after spinal anesthesia.
stroke index, expressed in ml/m2, is the ratio of stroke volume to the body surface area. | 30 min
  parameter will be measured using impedance cardiography and recorded every 5 min after spinal anesthesia.
systemic vascular resistance, expressed in Dynes.sec.cm-⁵ | 30 min
  parameter will be measured using impedance cardiography and recorded every 5 min after spinal anesthesia.
systemic vascular resistance index, expressed in Dynes.sec.cm-⁵/m2, is the ratio of systemic vascular resistance to the body surface area. | 30 min
  parameter will be measured using impedance cardiography and recorded every 5 min after spinal anesthesia.
stroke volume variation, expressed in percentage (%) | 30 min
  parameter will be measured using impedance cardiography and recorded every 5 min after spinal anesthesia.
systemic oxygen delivery, expressed in ml/min | 30 min
  parameter will be measured using impedance cardiography and recorded every 5 min after spinal anesthesia.
oxygen saturation, expressed in percentage (%) | 30 min
  parameter will be measured using pulse oximetry and recorded every 5 min after spinal anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Rafał Kowalczyk, PhD, Principal Investigator — I Department of Anaesthesiology and Intensive Care, Infant Jesus Teaching Hospital
Locations (1):
- Infant Jesus Teaching Hospital, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Primary and secondary outcomes will be available

REFERENCES:
- [Background] Abbasivash R, Sane S, Golmohammadi M, Shokuhi S, Toosi FD. Comparing prophylactic effect of phenylephrine and ephedrine on hypotension during spinal anesthesia for hip fracture surgery. Adv Biomed Res. 2016 Oct 26;5:167. doi: 10.4103/2277-9175.190943. eCollection 2016. PMID 27995106